CLINICAL TRIAL: NCT06717854
Title: Retrograde and Antegrade Enema for Prevention of Low Anterior Resection Syndrome After Low Anterior Resection: a Single-Center, Prospective Randomized Controlled Trial
Brief Title: Retrograde and Antegrade Enema for Prevention of LARS After LAR: a Randomized Controlled Trial
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sichuan Cancer Hospital and Research Institute (Other)
Responsible Party: Principal Investigator, Hui Yang, Principal Investigator, Sichuan Cancer Hospital and Research Institute
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: SCCHEC-02-2024-226
Record Dates: First submitted 2024-11-30; First posted 2024-12-05 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2024-11

CONDITIONS: Low Anterior Resection Syndrome
MeSH Terms: conditions — Low Anterior Resection Syndrome

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- standard of care (No Intervention): The standard of care (SOC) was implemented following low anterior resection, which included the distribution of pamphlets and instructional videos to patients and their caregivers.
- antegrade enema (Experimental): Participants assigned to this group received the standardized of care as the basis for the intervention. The enema is administered through the distal end of the ileocecal stoma, directed towards the anus.
- retrograde enema (Experimental): Participants assigned to this group received the standardized of care as the basis for the intervention. The enema is administered retrogradely via the anus.
  Interventions: Other: transanal irrigation

INTERVENTIONS:
Other: transanal irrigation — The enema is administered retrogradely via the anus. The enema commences one month post-operatively for patients with well-healed wounds, absence of stoma-related complications, and no evidence of anastomotic leakage upon digital examination, until ileostomy reversal. the catheter is gently and slowly inserted 7-10 cm through the anus. The initial irrigation volume is set at 500 ml and is gradually increased based on the patient's tolerance, up to a maximum of 1000 ml. 39-41°C warm water is the choice. Enemas are administered twice weekly, with each session limited to a duration of 30 minutes.
  Arms: retrograde enema
Other: antegrade enema — The enema is administered through the distal end of the ileocecal stoma, directed towards the anus. The enema commences one month post-operatively for patients with well-healed wounds, absence of stoma-related complications, and no evidence of anastomotic leakage upon digital examination, until ileostomy reversal. Using a disposable catheter, insert it about 20 cm. The initial irrigation volume is set at 500 ml and is gradually increased based on the patient's tolerance, up to a maximum of 1000 ml. 39-41°C warm water is the choice. Enemas are administered twice weekly, with each session limited to a duration of 30 minutes.

SUMMARY:
The goal of this clinical trial is to learn if enema works to prevent low anterior resection syndrome (LARS) in adults. The main questions it aims to answer are:

1. To describe the level of stoma adaptation before and after the patients received enemas during the stoma period as well as the levels and trends of LARS, bowel function, sleep quality, and quality of life after stoma reduction surgery
2. To compare the effects and advantages and disadvantages of antegrade and retrograde enema, and to investigate whether these two types of enema can provide safe and effective preventive measures for the prevention of LARS, the improvement of bowel function, and the enhancement of sleep and quality of life in rectal cancer patients after low anterior resection.

Researchers will compare antegrade enema, retrograde enema, and the standard of care to see if these two types of enema work to prevent LARS.

Participants will:

1. Receive either antegrade or retrograde enema or no enema based on the standard of care at 1 month after anterior rectal resection, until the ileostomy reversal.
2. Keep a diary of their symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Based on the NCCN guidelines for the pathological diagnosis of rectal cancer, patients are identified as having Primary Rectal Adenocarcinoma.
* ≥18 years.
* For the first time, anterior rectal dissection combined with prophylactic ileostomy was performed using laparoscopic, robotic, and open techniques.
* The patient exhibits normal cognitive and expressive abilities.
* Informed consent was obtained for voluntary participation in the study.

Exclusion Criteria:

* American Society of Anesthesiologists (ASA) Class III or higher.
* A combination of other intestinal conditions, including inflammatory bowel disease and Crohn's disease.
* Mental disorders and prolonged use of psychotropic medications.
* The presence of contraindications to enema administration.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2025-03-25 (Estimated); Primary Completion 2026-12-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
low anterior resection syndrome score (LARS score) | Pre-discharge, 1 month, 2 months, 3 months, 6 months after ileostomy reversal

SECONDARY OUTCOMES:
bowel function | before anterior rectal resection; 1 month, 2 months, 3 months, 6 months after stoma reversal
  Memorial Sloan Kettering Cancer Centre Bowel Function Instrument (MSKCC BFI)
quality of life for rectal cancer patients | before anterior rectal resection; 1 month, 2 months, 3 months, 6 months after stoma reversal
  quality of life will be measured using the EORTC Colorectal Cancer Module QLQ-CR29 (EORTC QLQ-CR29 )
quality of sleep | before anterior rectal resection, before starting enemas 1 month postoperatively, 2 months, 3-4 months postoperatively; 1 month, 2 months, 3 months, 6 months after stoma reduction
  Pittsburgh Quality Index (PSQI)

OTHER OUTCOMES:
Ostomy Adjustment Inventory-20 (OAI-20) | 1 month after anterior rectal resection before starting enemas, 2 months and 3-4 months postoperatively
A quality of life questionnaire for people with an ostomy (Stoma-QoL) | 1 month after anterior rectal resection before starting enemas, 2 months and 3-4 months postoperatively
Anal drainage and irritation during ileostomy (self-made) | 1 month after anterior rectal resection before starting enemas, 2 months and 3-4 months postoperatively

CONTACTS AND LOCATIONS:
Locations (1):
- Sichuan Clinical Research Center for Cancer, Sichuan Cancer Hospital & Institute, Sichuan Cancer Center, Afffliated Cancer Hospital of University of Electronic Science and Technology of China, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: Undecided